CLINICAL TRIAL: NCT02800694
Title: Role of the Single-shot Spinal Analgesia to Control Labour Pain in Appropriately-selected Primiparous Parturients: A Prospective Study
Brief Title: Role of the Single-shot Spinal Analgesia to Control Labour Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Collaborators: Dr Wegdan Ali Abdelrahman (Unknown); Dr Haidy Salah (Unknown)
Responsible Party: Principal Investigator, Ahmed Rabie Abdelraheim, Dr Ahmed Rabie Abdelraheim, lecturer of Obstetrics And Gynaecology, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUH2496
Record Dates: First submitted 2016-05-31; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Labour Analgesia
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: "bupivacainediluted with 1 ml of normal saline" and "25 μg fentanyl " — The intrathecal medication included 1ml of 0.5% heavy bupivacaine (5 mg) diluted with 1 ml of normal saline and 25 μg fentanyl. Then, the parturients were placed in the supine position with left lateral displacement produced by placing a wedge under the right hip to prevent aortocaval compression and hypotension. Supplemental oxygen was applied using nasal cannula (2-4 L/min). Routine monitoring included maternal vital signs, uterine contractions and fetal heart rate tracing. The cardiotocogram was recorded continuously throughout the study period

SUMMARY:
Labor pain is the most severe pain most women will endure in their lifetimes. The most complete and effective method of pain relief during childbirth is neuraxial labor analgesia which provides adequate analgesia without maternal or fetal sedation. Epidural and combined spinal-epidural (CSE) analgesia are the standard techniques performed in the developed countries. Having an epidural catheter in place produces flexibility with labor management. The catheter can be dosed intermittently for parturients in whom labor is prolonged, who require surgical manipulation for vaginal delivery, or who require cesarean section for delivery (1). However, unavailability of full-time epidural services in low-resource countries results in minimal or no analgesia provided to laboring parturients. The suitability of single-shot spinal analgesia has been previously studied in advanced, rapidly progressing labor in primiparous and multiparous women and was found that it may be a useful alternative for painless labor in the case of limited resources for epidural analgesia (2,3,4). However, duration of action is a limiting factor of intrathecal analgesia, particularly for primiparous women.

A 25 μg dose of fentanyl lasts 60-90 minutes. The study investigating the dose response relation for intrathecal fentanyl showed that the maximal analgesic effect is achieved at about 25 μg fentanyl. Above this dose, the duration of action increases but with increasing the incidence of side effects (5). Synergy has been noted between 25 μg of fentanyl and 2.5 mg of bupivacaine with analgesia lasting about 3 hours (6). The investigators hypothesized that increasing the bupivacaine dose to 5 mg with 25 μg fentanyl can prolong the duration of analgesia. So, this dosage combination can be used at an early stage in appropriately-selected primigravida parturients. The purpose of this study is to investigate the safety and effectiveness of single-dose spinal analgesia to control labor pain in properly-selected primiparous women in a tertiary referral maternity hospital

DETAILED DESCRIPTION:
This prospective study will be conducted in El-Minia Maternity University Hospital after obtaining approval from the hospital ethical committee and informed consent from the participating parturients. The study will be conducted in the period from July to october 2016. Candidates for spinal analgesia included primigravida parturients with ASA physical status I and II, term pregnancy of singleton fetus, all vertex presentation and uncomplicated pregnancies. Excluded from the study were patients with contraindications to regional anesthesia, diagnosed fetal abnormalities, allergy to the study drugs or previous systemic opioid administration. After the parturients being in active labor, dilated at least 4 to 5 cm and asking for painless labor, they were selected by an experienced obstetrician to receive spinal analgesia, based on obstetric parameters such as cervical dilatation and effacement and position of the fetal head.

Following monitoring with noninvasive blood pressure, electrocardiogram and pulse oximeter and recording of baseline vital signs, 18-G intravenous cannula was inserted and Ringer's solution 10 ml/kg was administered. Under strict aseptic technique, spinal analgesia was performed using pencil-point 25G spinal needle at the L3-L4 or L4-L5 interspace with the patients in the sitting position. The intrathecal medication included 1ml of 0.5% heavy bupivacaine (5 mg) diluted with 1 ml of normal saline and 25 μg fentanyl. Then, the parturients were placed in the supine position with left lateral displacement produced by placing a wedge under the right hip to prevent aortocaval compression and hypotension. Supplemental oxygen was applied using nasal cannula (2-4 L/min). Routine monitoring included maternal vital signs, uterine contractions and fetal heart rate tracing. The cardiotocogram was recorded continuously throughout the study period

ELIGIBILITY:
Inclusion Criteria:

* primigravida parturients with ASA physical status I and II, term pregnancy of singleton fetus, all vertex presentation and uncomplicated pregnancies.

After the parturients being in active labor, dilated at least 4 to 5 cm and asking for painless labor, they were selected by an experienced obstetrician to receive spinal analgesia, based on obstetric parameters such as cervical dilatation and effacement and position of the fetal head

Exclusion Criteria:

* patients with contraindications to regional anesthesia, diagnosed fetal abnormalities, allergy to the study drugs or previous systemic opioid administration

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-10 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) for assessment of degree of labour pain after administration of spinal analgesia | 6 hours after administration of spinal analgesia
Number of participants with treatment-related adverse events | Up to 24 hours after administration of spinal analgesia
Duration of pain relief | 12 hours after spinal analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed R Abdelraheim, MD, MRCOG, Principal Investigator — Department of Obstetrics and Gynaecology
Locations (1):
- Department of Obstetrics and Gynaecology, Minia University Hospital, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No